CLINICAL TRIAL: NCT06841757
Title: Efficacy of Remote Ischemic Preconditioning on Diastolic Function in Coronary Artery Bypass Surgery: A Randomized Controlled Study Comparing Diabetic and Non-Diabetic Patients
Brief Title: The Effect of Remote Ischemic Preconditioning on Diastolic Function in Coronary Artery Bypass Surgery Between Diabetic and Non-Diabetic Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alzahraa Khalil Marie (Other)
Responsible Party: Sponsor-Investigator, Alzahraa Khalil Marie, Assistant lecturer in Cairo university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-342-2024
Record Dates: First submitted 2025-02-13; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus; Diastolic Function
Keywords: Coronary artery bypass surgery; Diastolic function; Remote ischemic preconditioning
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diabetic with Remote ischemic preconditioning (Experimental): Remote Ischemic Preconditioning (RIPC) Patients will undergo Remote Ischemic Preconditioning using a blood pressure cuff inflated on the upper limb to induce ischemia and reperfusion, 40 mmHg above systolic pressure. The procedure will involve 3 cycles of inflation (5 minutes each) and deflation (5 minutes each) post intubation.
  Interventions: Behavioral: Remote ischemic preconditioning
- Non diabetic with Remote ischemic preconditioning (Experimental): Remote Ischemic Preconditioning (RIPC) Non-diabetic patients who undergo Remote ischemic preconditioning using the same ischemia/reperfusion protocol as the diabetic group.
  Interventions: Behavioral: Remote ischemic preconditioning
- Diabetic without Remote ischemic preconditioning (No Intervention): Diabetic patients who receive standard care for CABG surgery without Remote ischemic preconditioning
- Non diabetic without Remote ischemic preconditioning (No Intervention): Non-diabetic patients who receive standard care for CABG surgery without RIPC.

INTERVENTIONS:
Behavioral: Remote ischemic preconditioning — Patients will undergo Remote Ischemic Preconditioning using a blood pressure cuff inflated on the upper limb to induce ischemia and reperfusion, 40 mmHg above systolic pressure. The procedure will involve 3 cycles of inflation (5 minutes each) and deflation (5 minutes each) post intubation
  Arms: Diabetic with Remote ischemic preconditioning; Non diabetic with Remote ischemic preconditioning

SUMMARY:
This randomized controlled study aims to evaluate the effects of Remote Ischemic Preconditioning (RIPC) on diastolic function in patients undergoing coronary artery bypass grafting (CABG). The study will compare diabetic and non-diabetic patients to determine whether RIPC improves myocardial relaxation and reduces diastolic dysfunction, as assessed by the E/e' ratio at multiple time points during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled for elective isolated on-pump CABG surgery for two- to three-vessel coronary artery disease.
* Both males and females will be included.
* In the diabetic groups: Type II diabetes currently requiring and adhering to insulin therapy for at least the past 3 months
* During cardiopulmonary bypass, the temperature will range from 28-33°C using an esophageal temperature probe.
* Antegrade warm cardioplegia will be given by the cardiovascular perfusionist.
* Baseline diastolic function will be obtained preoperatively using transthoracic echocardiography done within the six months prior to the surgery

Exclusion Criteria:

* Combined CABG and valve surgery, emergency CABG.
* Type I diabetes, Type 2 diabetes managed with oral hypoglycemic agents without insulin in the past 3 months
* Peripheral vascular disease (PVD) affecting the upper limbs.
* Acute coronary syndrome (ACS); acute or recent myocardial infarction.
* Left ventricular ejection fraction ≤30%.
* Serious pulmonary disease necessitating oxygen supplementation or mechanical ventilation.
* Renal failure, defined as eGFR < 30 mL/min/1.73 m² or requiring renal replacement therapy (dialysis).
* Liver failure, including Child-Pugh Class B or C cirrhosis, severe hepatocellular dysfunction, or listed for liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
E/e' Ratio (Diastolic Function) | T1: immediately after anesthesia induction and intubation (baseline) T2: Immediately before cardiopulmonary bypass (CPB) T3: 10 minutes after reperfusion and separation from CPB T4: 45 minutes after separation from CPB and before transfer to the ICU
  Echocardiography (Tissue Doppler Imaging) will be used to measure the E/e' ratio, a reliable parameter for assessing left ventricular filling pressure and diastolic function. This is the primary method to evaluate the effect of Remote Ischemic Preconditioning (RIPC) on diastolic function in both diabetic and non-diabetic patients undergoing CABG.

SECONDARY OUTCOMES:
Mitral Inflow Velocities(E/A Ratio) | T1: immediately after anesthesia induction and intubation (baseline) T2: Immediately before cardiopulmonary bypass (CPB) T3: 10 minutes after reperfusion and separation from CPB T4: 45 minutes after separation from CPB and before transfer to the ICU
  Using TEE to measure E/A ratio
Deceleration Time (DT) | T1: immediately after anesthesia induction and intubation (baseline) T2: Immediately before cardiopulmonary bypass (CPB) T3: 10 minutes after reperfusion and separation from CPB T4: 45 minutes after separation from CPB and before transfer to the ICU
Cardiac Troponin Levels | Evaluate cardiac troponin levels postoperatively after 24 hours as a marker of myocardial injury
Systolic and diastolic Blood pressure | T1: immediately after anesthesia induction and intubation (baseline) T2: Immediately before cardiopulmonary bypass (CPB) T3: 10 minutes after reperfusion and separation from CPB T4: 45 minutes after separation from CPB and before transfer to the ICU
Inotropic Support: | During surgery
  Usage and dose.
LVEF | Compare between start and end of surgery
  Ejection fraction

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Alagaty Ehsan Alagaty, Professor of anesthesia, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175